CLINICAL TRIAL: NCT07341074
Title: BRAin INjury REcovery After Symptom-guided Early Therapy
Brief Title: Multicenter Early Intervention Study in Adults With Complaints After Mild Traumatic Brain Injury
Acronym: BRAIN-RESET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL-010193; 10390032310049 (Other Grant/Funding Number: ZonMW)
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment by physical- and or occupational therapist (Experimental)
  Interventions: Other: Treatment by physical- and/or occupational therapist
- Psychoeducation via telephonic counseling (Experimental)
  Interventions: Behavioral: Psychoeducation via telephonic counselling
- Care as usual (No Intervention)

INTERVENTIONS:
Other: Treatment by physical- and/or occupational therapist — Patients that are randomized in intervention arm 1 (physical- or occupational therapy) will be allocated for treatment by a physical therapist if the complaints are in the somatic domain, by an occupational therapist if the complaints are in the cognitive domain, and by both if the complaints are in both domains.
  Arms: Treatment by physical- and or occupational therapist
Behavioral: Psychoeducation via telephonic counselling — Patients randomised to the psychoeducation arm will be contacted by a research nurse by telephone three times between weeks 3 and 6 post-injury (approximately once per week). During the sessions, the patient's current symptoms, the expected course of recovery, and the overall favourable prognosis will be discussed based on a standardized telephone script. Reassuring information and general guidance will be provided, without the intention of inducing major behavioural change.
  Arms: Psychoeducation via telephonic counseling

SUMMARY:
Rationale: In the Netherlands, traumatic brain injury (TBI) is one of the most frequent neurological diseases and one of the leading causes of disability. Presumably, about half of the total Dutch population will get a TBI during their lifetime. The majority, about 85%, of patients suffers from a mild TBI (mTBI). The incidence of mTBI is estimated at 68,000 patients each year, but this is an underestimation as patients seen at the general practitioner's offices are not taken into account. In general, the prognosis of mTBI is relatively good, however more than 70% of patient still have one or more post-traumatic complaints at six months post-injury influencing resumption of daily (social) activities and return to work/study. Considering the high annual incidence of mTBI the number of patients with incomplete recovery has high social impact accompanied with excessive health care related costs. Post-traumatic complaints in the chronic phase postinjury are considered therapy resistant and so far no evidence based treatment is available. Hence, the most appropriate strategy is to prevent complaints present in the (sub)acute phase after injury to become persistent to improve functional outcome and quality of life.

Objective: The main aim of this study is to improve early care for patients suffering from post-traumatic complaints after mTBI through the development of effective symptom-guided tailored interventions. Nowadays, no effective therapy is available and care-as-usual consists of a wait-and-see policy. Early therapy will reduce posttraumatic complaints and facilitate earlier return to daily activities and work or study, consequently quality of life will be improved as well. This in turn will result in less healthcare consumption and lower societal costs.

Study design: The investigators propose a prospective three-arm multicenter open randomized controlled trial (RCT), randomizing participants between two interventions and care as usual. The end-point assessment is blinded.

Study population: Adults, aged 18-70 years, diagnosed with a mTBI at the Emergency Department (ED) of the participating hospitals within 24 hours after injury are eligible for inclusion.

Intervention: At two weeks post-injury the presence, severity, and type of post-traumatic complaints are assessed using the Rivermead Postconcussive complaints Questionnaire (RPQ). If a predefined minimum of complaints is present, a participant is randomised for one of the two interventions or the control group. The first intervention arm consists of symptom-targeted treatment with assignment to physical and/or occupational therapy. The second intervention arm involves psychoeducation about the complaints through telephonic counselling. The interventions are offered during three weeks from week 3-6 week post-injury.

Main study parameters/endpoints: The primary outcome measure is the total RPQ sum score at three months postinjury. The secondary outcome measures are functional outcome and quality of life.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants included in treatment arm 1 will undergo three to six therapy sessions with a physiotherapist and/or occupational therapist over a period of three weeks. This regimen may be potentially burdensome by its frequency but the risks associated with these treatments are low. Participants randomised to treatment arm 2 will receive three telephone calls over the course of three weeks, during which psychoeducation will be provided. This intervention is minimally burdensome and risk-free. All participants included in the interventional part of the study will complete questionnaires at three time points after injury and will receive two follow-up telephone calls three and six months post-injury for outcome assessment. This process is minimally burdensome and poses no risk. Finally, participants included in the registry will complete a limited set of questionnaires at three time points, which is also minimally burdensome and riskfree.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Seen at the ED within 24 hours after trauma
* Loss of consciousness (<30min.)
* Post-traumatic amnesia (<24hrs)
* Glasgow Coma Scale (GCS) score of 13-15 after initial resuscitation at the ED
* Comprehension of Dutch language

Exclusion Criteria:

* Inability for follow-up
* Chronic substance abuse (alcohol and/or drugs)
* Severe psychiatric disease
* Documented previous traumatic brain injury for which the patient was admitted
* Dementia and/or other severe comorbidities
* Current treatment by physical and/or occupational therapist for other indications
* Language barriers or illiteracy prohibiting understanding and completion of questionnaires

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic complaints (measured by Rivermead Post-concussion symptoms Questionnaire, RPQ) | Three months post-injury
  The RPQ is a validated questionnaire with sixteen questions assessing the presence and severity of post-traumatic complaints across somatic, cognitive, and emotional domains within the preceding 24 hours, in comparison to their pre-injury state. Responses are assigned on an ordinal scale from 0 to 4, with 0 indicating the absence of the complaint and 4 indicating a severe symptom.